CLINICAL TRIAL: NCT02056691
Title: Clinical and Biological Effects of a Preoperative Exercise Programme in Colorectal Tumour and Skeletal Muscle Tissues (Exercise inDuced Changes In Colorectal Cancer Tissues)
Brief Title: EDICT - Exercise inDuced Changes In Colorectal Cancer Tissues
Acronym: EDICT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Bournemouth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ed-1
Record Dates: First submitted 2014-02-05; First posted 2014-02-06 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Cancer
Keywords: Resectable; non-metastatic; colorectal; carcinoma; cancer; neoplasm; exercise; effects; program; pre-operative; proliferation; diagnosed; surgery; biopsy; muscle; signalling; IGF1; ki67; p53; response; training; biochemical; pathways; glucose
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma; Neoplasms; Motor Activity; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise programme (Experimental): Exercise programme Muscle biopsies
  Interventions: Procedure: Exercise programme; Procedure: Muscle biopsy

INTERVENTIONS:
Procedure: Exercise programme — The exercise regime consists of 10 sessions of exercise against a constant load, each lasting 60 seconds, separated by 60 seconds of recovery eliciting 90% maximal heart rate. The 6 sessions are held over a 2 week period.
Procedure: Muscle biopsy — muscle biopsy under local anaesthetic taken from the thigh, again for analysis and storage 3 times: before, during and after the exercise programme

SUMMARY:
This pilot study looks to explore the biological effects of exercise on cancer and muscle cells using a two week exercise program (HIThigh intensity training) on 20 patients with newly diagnosed and operable colorectal cancer following diagnosis and prior to surgery. Maximal oxygen uptake will also be measured. The aim of this pilot is to assess the feasibility of recruiting participants to and carrying out a two week preoperative exercise program in patients with colorectal cancer.

DETAILED DESCRIPTION:
Patients undergoing investigation for symptoms of colorectal cancer presenting to the hospital will undergo standard diagnostic procedures. Once resectable nonmetastatic cancer has been diagnosed (i.e. cancer that has not spread beyond the bowel), is amenable to surgical resection as decided by the colorectal multidisciplinary and if the patient fulfills the selection criteria, they will be asked if they wish to participate in the study. They will be given information regarding the study at the time of diagnosis. If they give their consent then a formal consenting process will take place at the next routine appointment.

During this appointment the patient will have the opportunity to ask questions. A member of the study team will explain the study in detail, answer any questions potential participants (and their partners/ carers) have. The patient is free to refuse participation or withdraw from the study at any time without this affecting their care, this is explained in the information and will be discussed further at the time of informed consent. If the patient agrees to participate in the trial, following the provision of informed consent and before embarking on the exercise programme they will need to fill in two questionnaires, the International Physical Activity Questionnaire (Long) and Dietary Intervention in Primary Care Questionnaire (DINE). They will be counseled to try and maintain their normal exercise level and their calorie intake. Blood samples will also be taken, analyzed and stored for further analysis including possible genetic analysis at a later stage before starting the exercise regime. They will have a muscle biopsy under local anaesthetic taken from the thigh, again for analysis and storage.

Participants will undergo an initial assessment of their baseline exercise ability and oxygen absorption using an upright exercise bike with concurrent ECG readings and breath analysis. The two week preoperative exercise regime will be planned depending on the patient's operation date. The exercise regime consists of 10 sessions of exercise against a constant load, each lasting 60s, separated by 60s of recovery eliciting 90% maximal heart rate.

The 6 sessions are held over a 2 week period. Each patients exercise ability and oxygen absorption will be remeasured at the end of the 2 week period and a second sample of blood taken for comparison. During the operation a sample of adipose tissue near the tumour site will be taken separately to the main sample. A muscle biopsy from the thigh will also be taken at the same time. As a standard of clinical care all patients are reviewed in the outpatient setting 6 weeks postoperatively. When patients attend this follow up appointment a final blood test and muscle biopsy (under local anaesthetic) will be taken to assess the longer term effects of the exercise program. Patient consent will be sought for this separately although it will be discussed at the initial introduction to the study.

Patients are free to withdraw from the study at any time and if there are any adverse events or concerns regarding the continuation of the study for a patient then they will be withdrawn.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer confirmed by histology
* Considered fit for surgery by surgical and anaesthetic team
* Considered fit for physical activity programme by MDT
* Age ≥ 18 years
* BMI ≥ 26 kg/m2
* Not pregnant
* Non obstructing cancer
* Able to provide written informed consent
* Patients not having neoadjuvant chemotherapy

Exclusion Criteria:

* Receiving hormone therapy
* Patients with diabetes
* Patients currently on either a dietary or exercise programme reflective of the World Cancer Research Fund Guidelines.
* Cardiac or renal impairment
* Excessive use of laxatives
* History of eating disorders
* Patients with inflammatory bowel disorders/coeliac
* Strong family history/polyposis (i.e. more than one 1st degree relative <55yrs)
* Patients with previous or concurrent malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10; Primary Completion 2017-09-19 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Assess the feasibility of carrying out a two week preoperative exercise program in patients with colorectal cancer and assess the effects of preoperative exercise on the proliferation of colorectal cancer cells | 1 year
  To assess the feasibility of carrying out a two week preoperative exercise program in patients with colorectal cancer and to assess the effects of preoperative exercise on the proliferation of colorectal cancer cells by measuring the change in the percentage of cells staining positive for Ki67 (a measure of cell proliferation).

SECONDARY OUTCOMES:
Changes in molecular markers for the effects of exercise and/or diet on AMPK/ mammilian target of rapamycin signalling pathway | 12 weeks
  Measuring changes in molecular markers for the effects of exercise and/or diet on AMPK/mTOR signalling pathway (phosphorylated 4EBP1 (P4EBP1), phosphorylated protein kinase B (PPKB/AKT), and phosphorylated AMPK (PAMPK).
Changes in AKT expression normal colonic tissue | 12 weeks
  Measuring changes in AKT expression normal colonic tissue - Intensity of AKT1/AKT2 staining, or AKT phosphorylation, a marker of insulin receptor signalling in cells.
Assessing Apoptosis index | 12 weeks
  Assessing Apoptosis index - Percentage of tumour cells staining positive for DNA fragmentation, a marker of cells undergoing apoptosis and therefore cell death.
Changes in molecular markers that may mediate or modify exercise/dietary effects in tumour tissues | 12 weeks
  Measuring changes in molecular markers that may mediate or modify exercise/dietary effects in tumour tissues (IR, IGF1R, p53 and its transcriptional target p21, ER, progesterone receptor, tumor necrosis factor-alpha converting enzyme and TIMP3).
Assessing gene expression profiles | 12 weeks
  Assessing gene expression profiles focusing on gene associated with insulin resistance.
Assessing the 11 gene signature | 12 weeks
  Assessing the 11 gene signature that help to predict maximal oxygen uptake gain in patients before and after exercise
Blood methylation profiles. | 12 weeks
  Blood methylation profiles.
Cortisol levels | 12 weeks
  Cortisol levels to evaluate levels of biological stress.
Postoperative complications up to 30 days postoperatively | 30 days post op
  Postoperative complications up to 30 days postoperatively
Moderator variables | 12 weeks
  Moderator variables including state of motivational readiness for exercise, weight change, depression and anxiety
Irisin levels | 12 weeks
  Irisin levels before and after exercise

CONTACTS AND LOCATIONS:
Overall Officials: Tamas Hickish, FRCP, Principal Investigator — The Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - The Royal Bournemouth Hospital, Bournemouth, Dorset
  - Poole Hospital, Poole, Dorset